CLINICAL TRIAL: NCT04013074
Title: Efficacy and Safety of Early TIPS (Transjugular Intrahepatic Portosystemic Shunts) in the Management of Cirrhosis With Recurrent Ascites.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-23
Record Dates: First submitted 2019-07-07; First posted 2019-07-09 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Liver Cirrhoses
MeSH Terms: interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIPS+Standard Medical Treatment (Experimental): TIPS along with standard medical therapy only included as per requirement nutritional therapy (high calorie intake- 2400 Kcal/ day) as and when required LVP and albumin infusion and diuretics.
  Interventions: Procedure: Transjugular Intrahepatic Portosystemic Shunt; Other: Standard Medical Treatment
- Standard Medical Treatment (Active Comparator): standard medical therapy only included as per requirement nutritional therapy (high calorie intake- 2400 Kcal/ day) as and when required LVP and albumin infusion and diuretics.
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Procedure: Transjugular Intrahepatic Portosystemic Shunt — Transjugular Intrahepatic Portosystemic Shunt
  Arms: TIPS+Standard Medical Treatment
Other: Standard Medical Treatment — Standard Medical Therapy only included as per requirement nutritional therapy (high calorie intake- 2400 Kcal/ day) as and when required LVP and albumin infusion and diuretics.

SUMMARY:
All consecutive patients with cirrhosis of liver who satisfy the criteria will be included and will be evaluated clinically along with all routine investigations and standard medical therapy will be continued among these patients. The patients between 18-60 yrs of age (cirrhosis diagnosed on the basis of clinical, biochemical, fibroscan & imaging.) , with ascites and HVPG (Hepatic Venous Pressure Gradient) >12, with 2 or more large volume paracentesis in last 3 month . CTP ≥ 7-13 will be considered for the study.

At baseline, a complete history of the cause of cirrhosis of liver with clinical and physical examination, a record of demographic profile, standard of care biochemical investigations would be done.

In this study patients who satisfy the inclusion and exclusion criteria as mentioned below will be enrolled to receive either standard medical therapy with Large volume paracentesis and albumin infusion or to be randomised to receive TIPS (Transjugular Intrahepatic Portosystemic Shunt).

The patients in group A will be given standard medical therapy only included as per requirement nutritional therapy (high calorie intake- 2400 Kcal/ day) as and when required Large Volume Paracentesis (LVP) and albumin infusion and diuretics.

ELIGIBILITY:
Inclusion Criteria:

1. Liver Cirrhotics between 18-60 yrs of age (cirrhosis diagnosed on the basis of clinical, biochemical, fibroscan & imaging)
2. Recurrent ascites (2 or more large volume paracentesis in last 3 month) on maximal tolerated diuretic dose.
3. Diuretic intractable ascites ( developing AKI/ hyponatremia (Na-<130 , hypo/ hyperkalemia (<3.5 , >5.5), who will respond to withdrawal of diuretics
4. HVPG >12 mm Hg
5. CTP ≥ 7-12
6. Patient is willing and able to comply with all study protocol requirements, including specified follow-up and testing.

Exclusion Criteria:

1. Hepatic or extra hepatic Malignancy-HCC, PVT
2. MELD (Model for End Stage Liver Disease) > 18
3. Post TIPS (Transjugular Intrahepatic Portosystemic Shunt), Shunt surgery
4. LVP (Large Volume Paracentesis) >3/month
5. Acute kidney injury (Sr.Cr>2mg/dl)

5) CKD (Chronic Kidney Injury) 6) Previous hepatic encephalopathy 7) Acute on chronic liver failure 8) Active infection 9) Active alcohol intake 10) Left Ventricular systolic dysfunction/ overt CCM 11) PPH (Portopulmonary Hypertension) 12) Pt on mechanical ventilation 13) Patient in ICU/ any acute illness 14) Pregnant lady 15) SBP (Spontaneous bacterial Peritonitis)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival in both groups | 1 year

SECONDARY OUTCOMES:
Overall survival in both groups | 1 year
Reduction in HVPG from baseline in both groups | 6 month
Reduction in HVPG from baseline in both groups | 12 month
Incidence of Acute Kidney Injury new complications in both groups | 1 year
Incidence of Spontaneous bacterial Peritonitis in both groups | 1 year
Incidence of Hepatic Encephalopathy in both groups | 1 year
Incidence of Bleeding in both groups | 1 year
Incidence of hyponatremia in both groups | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided